CLINICAL TRIAL: NCT02076191
Title: Multicenter Phase I/II Trial of Ruxolitinib in Combination With Decitabine in Patients With Accelerated Phase Myeloproliferative Neoplasm (MPN) or Post-MPN AML
Brief Title: Study of Combination Ruxolitinib and Decitabine Treatment for Accelerated Phase MPN or Post-MPN AML
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: John Mascarenhas (Other)
Collaborators: Myeloproliferative Disorders-Research Consortium (Network); National Cancer Institute (NCI) (NIH); Incyte Corporation (Industry)
Responsible Party: Sponsor-Investigator, John Mascarenhas, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 13-1816; MPD-RC 109 (Other: Myeloproliferative Disorders-Research Consortium); P01CA108671 (NIH)
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Myeloproliferative Neoplasms
Keywords: Ruxolitinib; Decitabine; Myeloproliferative Neoplasms; Combination Therapy
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — ruxolitinib; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Myeloproliferative neoplasms (Experimental): In phase I, increasing doses of ruxolitinib in combination with decitabine at a dose of 20 mg/m2 daily intravenously over 5 days. An initial dose of ruxolitinib of 10 mg orally twice daily is anticipated with planned, dose escalations of 15 mg orally twice daily, 25 mg orally twice daily and 50 mg orally twice daily. The dose can also be de-escalated to 5mg orally twice daily if dose limiting toxicities (DLTs) are observed at the initial 10mg dose. Patients will receive ruxolitinib as a single agent for the first 7 days followed by the administration of decitabine on day 8 for a total of 5 consecutive days. Patients will continue ruxolitinib at the assigned dose through the first cycle and may reduce the dose for specified toxicity beginning with the second cycle. Patients in Phase II will start at the recommended phase II dose (RPTD) of ruxolitinib in combination with decitabine at a dose of 20 mg/m2 daily intravenously over 5 days.
  Interventions: Drug: Ruxolitinib; Drug: Decitabine

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib will be administered at doses of 5mg, 10mg, 15mg, or 25 mg taken orally every 12 hours throughout the treatment cycle.
Drug: Decitabine — Decitabine is administered intravenously at a dose of 20 mg/m2 daily for 5 days. Subsequent cycles of decitabine may be administered at 4 week intervals as clinically tolerated. Decitabine treatment may be deferred for up to 2 weeks to allow recovery from non-hematologic toxicity during the first 6 cycles and up to 2 weeks thereafter for hematologic toxicities as well. The first treatment cycle will last 35 days and will be the evaluable period for DLTs and RPTD determination for patients enrolled in the phase I portion only. Subsequent treatment cycles will be 4-6 weeks in duration as defined by decitabine administration.

SUMMARY:
The purpose of this study is to test the safety and tolerability of ruxolitinib at different dose levels in combination with decitabine and the effectiveness of ruxolitinib in combination with decitabine in patients with accelerated or blast phase Myeloproliferative Neoplasm (MPN), which is a group of diseases of the bone marrow in which excess cells are produced. Ruxolitinib is a drug that is approved by the Federal Drug Administration (FDA) for the treatment of patients with advanced forms of myelofibrosis. It inhibits the Jak proteins that are often abnormal in MPN. A recent clinical study showed that ruxolitinib treatment could put some patients with this disease into remission. Decitabine is a chemotherapy, approved by the Federal Drug Administration (FDA), that has been used to treat acute leukemia. It works in some patients, but most patients with accelerated and blastic MPN do not respond to treatment. Ruxolitinib and decitabine will be combined in this study to find out what dose of the two medicines are safe together. Using Ruxolitinib in combination with Decitabine is experimental. The investigators want to find out what effects, good and/or bad it has on the patient and the disease.

DETAILED DESCRIPTION:
At this time, there is no standard medical treatment for MF-BP or MF-AP. The investigators believe that the combination of ruxolitinib and DEC is a candidate approach to the treatment of MF-BP/MF-AP that is worthy of exploration based on both the current understanding of the biology of disease and emerging preclinical data. The molecular pathogenesis of MPN and progression to blast phase is almost certainly due to a complex combination of gene mutations (JAK2V617F, MPL) and epigenetic alterations (IDH1/2, IKZF1, EZH2, TET2) that culminate in the emergence of leukemic clones. Recent evidence indicates that the JAK2V617F protein can localize in the nucleus and influence global DNA methylation patterns which may lead to genomic instability and disease progression. The inhibition of JAK-STAT mediated cell proliferation and survival in conjunction with the reversal of DNA hypermethylation of tumor suppressor genes would be predicted to have at least an additive if not synergistic effect in inducing apoptosis of cells belonging to the malignant myeloid clone. Correlative studies conducted within a trial of Private and Confidential MPD-RC 109 Ruxolitinib + Decitabine combination JAK2 inhibitor and DMNT1 inhibitor in patients with MPN-BP would explore the effect on methylation status of various gene promoters as well as the influence on gene expression of chromatin related proteins and ultimately leukemic cell survival. The sequential administration of a JAK2 inhibitor followed by a DNMT inhibitor would also potentially serve to overcome the JAK2-independent effects of epigenetic lesions that lead to MPN-BP. In addition, a murine model of leukemic transformation has been described. In this model, bone marrow obtained from Tp53 null mice is retrovirally transduced with Jak2V617F, and transplanted into donor C56BL/6 mice. The transplanted mice develop an MPN which progresses to AML. In vitro drug studies utilizing bone marrow from these leukemic mice have demonstrated that exposure to decitabine or ruxolitinib inhibits colony formation in a methylcellulose colony-forming assay. Importantly, the combination of decitabine and ruxolitinib in this assay significantly reduces colony formation when compared to either drug alone (Rampal et al. ASH 2012 oral abstract 808) thus providing pre-clinical evidence for the combination study proposed here.

ELIGIBILITY:
Inclusion Criteria:

* Accelerated phase MPN as defined by 10%-19% blasts in the peripheral blood or bone marrow and evidence of dysplastic marrow features with a concomitant diagnosis of essential thrombocythemia (ET), polycythemia vera (PV) or primary myelofibrosis (PMF) or a diagnosis of acute myelogenous leukemia as defined by 20% blasts in the blood or bone marrow following a previous diagnosis of ET, PV or PMF.
* >18 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0-2. Patients with ECOG performance status of 3 will be eligible if the lower performance status is deemed by the investigator to be due entirely to accelerated or blastic phase MPN and not due to another comorbidity.
* Acceptable pre-study organ function during screening as defined as: Total bilirubin < 1.5 times the upper limit of normal (ULN) unless due to Gilbert's disease or hemolysis, Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN, Serum creatinine ≤ 1.5 x ULN
* Women of childbearing potential and males must agree to use adequate contraception (i.e., hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a female subject become pregnant or suspect she is pregnant while participating in this study, she should inform the treating physician immediately.
* Patients who are not candidates for or have declined an allograft.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Have had chemotherapy or investigational therapy, with the exception of hydroxyurea, within 4 weeks of study entry. Previous treatment with either ruxolitinib or decitabine as single agents will not exclude eligibility. Previous stem cell transplant will also not exclude eligibility as long as other inclusion/exclusion criteria have been met.
* Patients with acute myelofibrosis are excluded.
* Uncontrolled intercurrent illness including, but not limited to hepatitis, human immunodeficiency virus (HIV)-positive subjects receiving combination antiretroviral therapy, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, ventricular arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Other medications, severe acute/chronic medical or psychiatric conditions, or laboratory abnormalities that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, that in the judgment of the Investigator would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-02; Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | up to 5 weeks
  Safety and efficacy of ruxolitinib when used in combination with decitabine. MTD is defined as the highest dose studied for which the incidence of (Dose Limiting Toxicities) DLT is at least 33%.
Dose Limiting Toxicities (DLT) | up to 5 weeks
  Safety and efficacy of ruxolitinib when used in combination with decitabine. DLTs will be defined as those adverse events occurring in the first 5 weeks after initiation of therapy that are not clearly related to disease.

SECONDARY OUTCOMES:
Recommended Phase II Dose (RPTD) | up to 20 weeks
  Safety and tolerability of drug combination of ruxolitinib and decitabine. RPTD is that dose level below the MTD for which the incidence of DLT is <33%.

CONTACTS AND LOCATIONS:
Overall Officials: John Mascarenhas, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Ronald Hoffman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (8):
- United States (8):
  - Washington University of St. Louis, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center Institute, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Mascarenhas JO, Rampal RK, Kosiorek HE, Bhave R, Hexner E, Wang ES, Gerds A, Abboud CN, Kremyanskaya M, Berenzon D, Odenike O, Farnoud N, Krishnan A, Weinberg RS, McGovern E, Salama ME, Najfeld V, Medina-Martinez JS, Arango Ossa JE, Levine MF, Zhou Y, Sandy L, Heaney ML, Levine RL, Mesa RA, Dueck AC, Hoffman R. Phase 2 study of ruxolitinib and decitabine in patients with myeloproliferative neoplasm in accelerated and blast phase. Blood Adv. 2020 Oct 27;4(20):5246-5256. doi: 10.1182/bloodadvances.2020002119. PMID 33104796